CLINICAL TRIAL: NCT06493695
Title: Cranial Electrical Stimulation and Exercise Group Chatbot
Brief Title: CES and EGChatbot in Reducing Anxiety, Depression, Insomnia, and Mental Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH113-REC3-050
Record Dates: First submitted 2024-06-23; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Depression, Anxiety
Keywords: At-Risk Mental State; Exercise Chatbot; Cranial Electrotherapy Stimulation; Cognitive Mental Risks; Emotional Distress; Anxiety; Depression; Insomnia; Quality of Life
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: a randomized controlled experimental design with three groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chatbot & CES (Experimental): Exercise Chatbot intervention with Cranial Electrical Stimulation intervention
  Interventions: Behavioral: Both EGChat and CES intervention
- Chatbot (Experimental): Exercise Chatbot intervention without Cranial Electrical Stimulation intervention
  Interventions: Other: Exercise Chatbot
- CES (Experimental): Cranial Electrical Stimulation intervention without Exercise Chatbot intervention
  Interventions: Device: CES (Cranial Electrotherapy Stimulation)

INTERVENTIONS:
Behavioral: Both EGChat and CES intervention — 1. A exercise-promoting chatbot called EGChat, integrated into an established online health promotion platform.
  2. Intervention of CES (Cranial Electrotherapy Stimulation) at Home
  Other Names: EGChat and CES intervention
  Arms: Chatbot & CES
Other: Exercise Chatbot — Exercise Chatbot
  Arms: Chatbot
Device: CES (Cranial Electrotherapy Stimulation) — Intervention of CES (Cranial Electrotherapy Stimulation)
  Arms: CES

SUMMARY:
The objective of this three-year study is to provide comprehensive care to young adults presenting with ARMS. The aim is use an exercise group (EGChat) developed by prior study and CES to decrease cognitive mental risks, improve emotional stability, enhance sleep quality, and elevate overall life satisfaction. A randomized controlled trial (RCT) design will be conducted using purposive sampling to recruit 180 young adults with ARMS from a medical center and its affiliated hospitals. Participants will be randomly assigned to one of three groups, undergoing a 16-week intervention: EGChat plus CES, EGChat without CES, or CES without EGChat groups. The study integrates the EGChat application into an online health promotion platform, coupled with CES intervention, to enhance the biological and psychological health of individuals at ARMS. The goal of this RCT study is to enhance the biological and psychological well-being of individuals with ARMS, covering exercise levels, Brain-Derived Neurotrophic Factor (BDNF) levels, health-promoting behaviors, metabolic indexes, cognitive mental risks, emotional status, sleep quality, and overall life quality. Assessments will occur at baseline (T0), 8 weeks into the intervention (T1), upon completion of the 16-week intervention (T2), and during a follow-up assessment at 3 months post-intervention (T3). The study will utilize generalized estimating equations (GEE) for mixed model repeated measures analysis to evaluate the significant influences of the intervention and interactions between study variables, utilizing group-time interaction.

DETAILED DESCRIPTION:
In our previous study, the two-year psychosis transition rate was 8.33%, comparatively lower than rates reported in other international studies. Our findings highlight that individuals in the at-risk mental state (ARMS) category face cognitive, emotional, and sleep-related challenges, leading to compromised self-identity and impairments in daily functioning. A significant proportion of young adults at risk of mental health issues not only display cognitive vulnerabilities but also endure emotional instability and sleep disturbances, increasing the likelihood of suicidal ideation and persistent self-harming behaviors. It's clear that individuals facing mental health challenges, especially those with ARMS, require support from the health system. Exercise has been linked to enhanced cognitive function and mental health. The mental health chatbot as a promising tool for adolescents and young adults in the ARMS, showing potential in alleviating anxiety, depression, and mental health risks. Additionally, cranial electrotherapy stimulation (CES) is recommended as a safe and effective approach to address sleep-related problems. Together, these interventions may be proposed as a comprehensive care strategy, providing secure support for individuals with ARMS.

The objective of this three-year study is to provide comprehensive care to young adults presenting with ARMS. The aim is use an exercise group (EGChat) developed by prior study and CES to decrease cognitive mental risks, improve emotional stability, enhance sleep quality, and elevate overall life satisfaction. A randomized controlled trial (RCT) design will be conducted using purposive sampling to recruit 180 young adults with ARMS from a medical center and its affiliated hospitals. Participants will be randomly assigned to one of three groups, undergoing a 16-week intervention: EGChat plus CES, EGChat without CES, or CES without EGChat groups. The study integrates the EGChat application into an online health promotion platform, coupled with CES intervention, to enhance the biological and psychological health of individuals at ARMS. The goal of this RCT study is to enhance the biological and psychological well-being of individuals with ARMS, covering exercise levels, Brain-Derived Neurotrophic Factor (BDNF) levels, health-promoting behaviors, metabolic indexes, cognitive mental risks, emotional status, sleep quality, and overall life quality. Assessments will occur at baseline (T0), 8 weeks into the intervention (T1), upon completion of the 16-week intervention (T2), and during a follow-up assessment at 3 months post-intervention (T3). The study will utilize generalized estimating equations (GEE) for mixed model repeated measures analysis to evaluate the significant influences of the intervention and interactions between study variables, utilizing group-time interaction. Additionally, a machine-learning framework for EGChat will be implemented to enhance outcome predictions. The analysis of these machine-learning algorithms will be conducted using the WEKA software.

Comprehensive care intervention programs for individuals with ARMS should address the management of cognitive mental risks, anxiety, depression, and insomnia. The study findings provide evidence supporting the effectiveness of EGChat and CES in assisting young adults with ARMS. The ultimate goals are to achieve early intervention, delay the onset of psychosis, impede disease progression, and enhance the patient's capacity for self-management and societal adaptation.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years old
* meet the DSM-5 criteria for ARMS as assessed by psychiatrists, who serve as the Co-PI of this research
* exhibit persistent symptoms without clinically significant fluctuations
* consent to participate in the study and provide written informed consent.

Exclusion Criteria:

* have a DSM-5 diagnosis of intellectual disability or substance (including alcohol) use disorder
* possess a history of epilepsy, head trauma, central nervous system diseases, or frequent syncope
* are pregnant or lactating
* have an implanted neurostimulator or cardiac pacemaker
* have metal implants in the body
* non-removable cochlear implant
* are unable to adhere to the protocol (including the absence of a computer, tablet, or smartphone for use)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Levels of Cognitive Mental risk | week 0 (before interventions), weeks 8 (in the middle of 16 weeks interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  Chinese Version of Schizotypal Personality Questionnaire-Brief (range from 0-114 scores) and Scale of Prodromal Symptoms (range from 0-22 scores)。Higher scores mean a higher cognitive risk.
Levels of State Anxiety and Trait Anxiety | week 0 (before interventions), weeks 8 (in the middle of 16 weeks interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  Chinese Mandarin State-Trait Anxiety Inventory Form Y (range from 40-160 scores)。Higher scores mean a higher anxiety levels.
Levels of Depression | week 0 (before interventions), weeks 8 (in the middle of 16 weeks interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  Taiwanese Depression Scale (range from 0-66 scores)。Higher scores mean a higher depression levels.
Levels of Sleep Quality | week 0 (before interventions), weeks 8 (in the middle of 16 weeks interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  Pittsburgh Sleep Quality Index (range from 0-21 scores)。Higher scores mean a worse sleep problems.
Levels of Health-Promoting Lifestyle | week 0 (before interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  Short Health-Promoting Lifestyle Profile checklist (range from 24-96 scores)。Higher scores mean a better health promotion lifestyle.
Number of participants with Incidence of metabolic indicators | week 0 (before interventions), weeks 8 (in the middle of 16 weeks interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  Metabolic and Physical Measures。Higher numbers of indicators mean a worse outcomes in metabolic health status.
Levels of Quality of Life Questionnaire | week 0 (before interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  World Health Organization Quality of Life Assessment (range from 28-140 scores)。Higher scores mean a better lif quality.
Levels of Exercise | week 0 (before interventions), weeks 16 (after interventions), 3 months follow-up (post intervention)
  3-Month Physical Activity Checklist (self-report) and Actigraphy (Objective measure)。Higher scores mean a higher exercise levels.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Ma, PHD, Principal Investigator — School of Nursing
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No